CLINICAL TRIAL: NCT03888105
Title: An Open-Label Study to Assess the Anti-Tumor Activity and Safety of REGN1979, an Anti-CD20 x Anti-CD3 Bispecific Antibody, in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A Study to Assess the Anti-Tumor Activity and Safety of Odronextamab in Adult Patients With B-cell Non-Hodgkin Lymphoma Who Have Been Previously Treated With Other Cancer Therapies
Acronym: ELM-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-ONC-1625; 2017-002139-41 (EudraCT Number); 2024-511747-25-00 (Registry Identifier: CTIS number)
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: B-cell Non-Hodgkin Lymphoma (B-NHL)
Keywords: Relapsed B-NHL; Refractory B-NHL; NHL; Follicular lymphoma (FL); Diffuse large B-cell lymphoma (DLBCL); Mantle cell lymphoma (MCL); Marginal zone lymphoma (MZL); bispecific antibody; CD20
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Intervention Model Description: 5 cohorts The first 68 patients in the DLBCL cohort will be randomized; the remaining patients will not be randomized
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- FL (Experimental): Follicular lymphoma grade 1-3a cohort
  Interventions: Drug: Odronextamab
- DLBCL (Experimental): Diffuse large B-cell lymphoma cohort
  Interventions: Drug: Odronextamab
- MCL (Experimental): Mantle Cell Lymphoma cohort
  Interventions: Drug: Odronextamab
- MZL (Experimental): Marginal Zone Lymphoma cohort
  Interventions: Drug: Odronextamab
- Other B-NHL (Experimental): Other B-cell non-Hodgkin lymphoma cohort (excluding FL Grade 1-3a, DLBCL, MCL, MZL, Waldenström macroglobulinemia [WM]); Patients with a current diagnosis of mixed histology of B-NHL with an aggressive component (such as concurrent FL and DLBCL) will be allowed
  Interventions: Drug: Odronextamab

INTERVENTIONS:
Drug: Odronextamab — Administered by intravenous (IV) infusion
  Other Names: REGN1979

SUMMARY:
This study is researching an investigational drug, odronextamab, in adult patients B-cell non-Hodgkin's lymphoma (B-NHL).

The main purpose of this study is to assess the effectiveness of odronextamab in destroying cancer cells and to learn more about the safety of odronextamab.

The study is looking at several other research questions, including:

* To see if odronextamab works to destroy cancer cells
* Side effects that may be experienced by people taking odronextamab
* How odronextamab works in the body
* How much odronextamab is present in the blood

ELIGIBILITY:
Key Inclusion Criteria:

1. For the FL grade 1-3a cohort only: Central histopathologic confirmation of the FL Grade 1 to 3a diagnosis must be obtained before study enrollment. Patients with FL grade 3b are ineligible for this cohort but may be included in the "other B-NHL" cohort. Follicular lymphoma subtyping is based on the World Health Organization (WHO) classification (Swerdlow, 2017)
2. Disease-specific cohorts:

   Patients should in the judgment of the investigator require systemic therapy for lymphoma at the time of study enrollment
   * FL grade 1-3a cohort: Patients with FL grade 1-3a that has relapsed after or is refractory to at least 2 prior lines of systemic therapy, as defined in the protocol
   * DLBCL cohort: Patients with DLBCL that has relapsed after or is refractory to at least 2 prior lines of systemic therapy as defined in the protocol
   * MCL after BTK inhibitor therapy cohort: Patients with MCL who have relapsed or refractory disease to at least one prior line of systemic therapy and had prior treatment with a Bruton's tyrosine kinase (BTK) inhibitor
   * MZL cohort: Patients with MZL that have relapsed or is refractory to at least 2 prior lines of systemic therapy
   * Other B-NHL cohort: Patients with B-NHL other than FL grade 1-3a, DLBCL, MCL, or MZL that has relapsed after or is refractory to at least 2 prior lines of systemic therapy as defined in the protocol. New enrollment stopped for patients with Burkitt lymphoma and Burkitt-like lymphoma.
3. Measurable disease on cross sectional imaging as defined in the protocol documented by diagnostic imaging (computed tomography (CT), or magnetic resonance imaging (MRI)
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
5. Adequate bone marrow, hepatic, and renal function as defined in the protocol

Key Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or known involvement by non-primary CNS Non-Hodgkin Lymphoma (NHL) (suspected CNS lymphoma should be evaluated by lumbar puncture, as appropriate, in addition to the mandatory head CT or MRI)
2. Treatment with any systemic anti-lymphoma therapy within 5 half-lives or within 28 days prior to first administration of study drug, whichever is shorter
3. History of allogeneic stem cell transplantation, up to 12 months prior to first administration of study drug. The presence of acute or chronic graft-versus host disease (GVHD) will also be an exclusion
4. Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone or anti-inflammatory equivalent within 72 hours of start of study drug
5. History of neurodegenerative condition or CNS movement disorder. Patients with a history of seizure within 12 months prior to study enrollment are excluded
6. Another malignancy except B-NHL in the past 5 years, with the exception of non-melanoma skin cancer that has undergone potentially curative therapy or in situ cervical carcinoma, or any other tumor that has been deemed to be effectively treated with definitive local control and with curative intent
7. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection; cytomegalovirus (CMV) infection as noted by detectable levels on a blood polymerase chain reaction (PCR) assay as defined in the protocol or other uncontrolled infections
8. Known hypersensitivity to both allopurinol and rasburicase
9. Prior treatment with an anti-CD20 x anti-CD3 bispecific therapy

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR), as assessed by independent central review | Up to 52 weeks of study treatment
  FL grade 1-3a/MZL
ORR, as assessed by independent central review | Up to 36 weeks of study treatment
  DLBCL/MCL/Other B-NHL

SECONDARY OUTCOMES:
ORR, as assessed by the local investigator | Up to 52 weeks of study treatment
  FL/MZL
ORR, as assessed by the local investigator | Up to 36 weeks of study treatment
  DLBCL/MCL/Other B-NHL
Complete Response (CR) Rate, as assessed by the local investigator | Up to 52 weeks of study treatment
  FL grade 1-3a/MZL
CR rate, as assessed by independent central review | Up to 52 weeks of study treatment
  FL grade 1-3a/MZL
CR rate, as assessed by the local investigator | Up to 36 weeks of study treatment
  DLBCL/MCL/Other B-NHL
CR rate, as assessed by independent central review | Up to 36 weeks of study treatment
  DLBCL/MCL/Other B-NHL
Progression-Free Survival (PFS), as assessed by independent central review | Approximately 194 weeks following the first dose
PFS, as assessed by the local investigator | Approximately 194 weeks following the first dose
Overall Survival (OS) | Approximately 194 weeks following the first dose
Duration Of Response (DOR), as assessed by independent central review | Approximately 194 weeks following the first dose
DOR, as assessed by the local investigator | Approximately 194 weeks following the first dose
Disease Control Rate (DCR), as assessed by independent central review | Up to 52 weeks of study treatment
  FL grade 1-3a/MZL
DCR, as assessed by the local investigator | Up to 52 weeks of study treatment
  FL grade 1-3a/MZL
DCR, as assessed by independent central review | Up to 36 weeks of study treatment
  DLBCL/MCL/Other B-NHL
DCR, as assessed by the local investigator | Up to 36 weeks of study treatment
  DLBCL/MCL/Other B-NHL
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) | Approximately 194 weeks following the first dose
Concentration of odronextamab | 12 weeks following end of treatment
  End of infusion [EOI]; Concentration at a specified time t [Ct])
Incidence of Anti-Drug Antibodies (ADA) to odronextamab over time | 12 weeks following end of treatment
Titer of anti-drug antibodies to odronextamab over time | 12 weeks following end of treatment
Incidence of Neutralizing antibodies (Nab) to odronextamab over time | 12 weeks following end of treatment
Changes in scores of patient-reported outcomes as measured by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Cancer-30 (EORTC-QLQ-C30) | Approximately 194 weeks following the first dose
  The EORTC QLQ-C30 is a self-reported, 30-item generic questionnaire developed to assess 15 domains: global health status scale, five functional scales (physical, role, emotional, cognitive, and social functioning) and nine symptom scales (fatigue, nausea, vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties).
Changes in scores of patient-reported outcomes as measured by Functional Assessment of Cancer Treatment-Lymphoma (FACT-Lym) | Approximately 194 weeks following the first dose
  Composed of the FACT-G plus the 15-item Lymphoma Subscale (LymS).
Changes in scores of patient-reported outcomes as measured by EuroQol-5 Dimensions-3 Levels (EQ-5D-3L) | Approximately 194 weeks following the first dose
  The EQ-5D-3L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (119):
- United States (13):
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Weill Cornell Medical College New York Presbyterian Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
- Australia (7):
  - Border Medical Oncology, East Albury, New South Wales
  - Northern NSW Local Health District The Tweed Hospital, Tweed Heads, South Wales
  - Epworth Hospital, East Melbourne, Victoria
  - North Building, Frankston, Victoria
  - Andrew Love Cancer Centre, Geelong, Victoria
  - Olivia Newton John Cancer Wellness & Research Centre, Heidelberg, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - QEII Health Science Centre - Halifax location, Halifax, Nova Scotia
- China (17):
  - Peking University Cancer Hospital (Beijing Cancer Hospital) (Beijing Institute for Cancer Research), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Beijing Municipality
  - Second Affiliated Hospital - Xinqiao Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-Sen University Cancer Center - Cancer Prevention and Treatment Center, Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Tumor Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital - Soochow University, Suzhou, Jiangsu
  - The First Bethune Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Shanhai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute, Tianjin, Tianjin Municipality
  - The First Hospital affiliated to the Medical School of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Peking University - Third Hospital, Beijing
- France (9):
  - Hopital Haut-Leveque, Pessac, Aquitaine
  - Centre Hospitalier Universitaire de Caen - Hematologie Clinique IHBN, Caen, Calvados
  - Hopital Lyon Sud, Pierre-Bénite, Lyon
  - Hopital Claude Huriez - CHR Lille, Lille, Nord
  - CHU Hotel Dieu Service Hematologie, Nantes, Pays de la Loire Region
  - Chu Poitiers - Pole Regional De Cancerologie, Poitiers, Vienne
  - Hopital Saint Louis, Paris
  - Hospital de la Pitie-Salpetriere, Paris
  - Unite Hemopathies Lymphoides Hospital Henri Mondor, Créteil, Île-de-France Region
- Germany (3):
  - Kliniken Ostalb Stauferklinikum Schwab Gmund, Mutlangen, Gmund
  - University Hospital Halle Saale, Halle
  - Universitatsklinik Wurzburg, Med Klinik und Poliklinik II, Zentrum Innere Medizin, Würzburg
- Italy (10):
  - UOC Hematologia, Fondazione IRCCS, Ca Granda, OM Policlinico, Milan, Milan
  - University of Bologna Dipartimento di Medicina Specialistica Diagnostica e Sperimentale, Bologna
  - Uos Ematologia - Ospedale Civile di Livorno, Livorno
  - ASST Grande Ospedale Metropolitano Niguarda - Division of Hematology, Milan
  - AOU Maggiore della Carita, Novara
  - Presidio Ospedaliero Santa Maria della Misericordia, Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale dell'Angelo - Varese, Varese
  - Ospedale DellAngelo Di Mestre, Venice
- Japan (14):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aiti
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization National Kyushu Cancer Center, Fukuoka, Hukuoka
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara-Shi, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Cancer Center Hospital - Tsukiji Campus, Chuo Ku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
- Poland (8):
  - Centrum Onkologii Instytut im M Sklodowskiej CurieOddzial Chorob United Kingdomladu Chlonnego, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum, Gdansk, Pomeranian Voivodeship
  - Pomorskie Hospitals SP. Z O. O. Oncology And Radiotherapy Ward, Gdynia, Pomeranian Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie spSp. Z.o.o., Gdynia
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. Mikolaja Kopernika w Lodzi (Copernicus Memorial Hospital), Lodz
  - Instytut Hematologii I Transfuzjologii Klinika Hematologii, Warsaw
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Klinika Hematologii, Terapii Komorkowych i Chorob Wewnetrznych, Wroclaw
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Icon Soc Farrer Park, Singapore
- South Korea (8):
  - University of Ulsan College of Medicine, Ulsan, Daegu
  - National Cancer Center, Gyeonggi-do, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Ewha Womans University Mokdong Hospital - Hemato Oncology, Seoul
- Spain (12):
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital Son Llatzer, Palma, Balearic Islands
  - Ico Lhospitalet - Hospital Duran i Reynals, Barcelona, Catalonia
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona - Planta 4 Escalera, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (8):
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - China Medical University, Taichung
  - National Cheng Kung University, Tainan
  - Chi-Mei Medical Center - Liuying, Tainan
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation-, Taoyuan District
- United Kingdom (5):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Derriford Hospital and the Royal Eye Infirmary, Plymouth, Devon
  - The Royal Marsden Hospital, Sutton, Surrey
  - University Hospital of Wales, Cardiff, Wales
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Arnason JE, Matasar M, Luminari S, Tucker D, Sun D, Tao W, Zhu YO, Kundu K, Gupta NT, Leary A, Jankovic V, Ambati S, Mohamed H, Chaudhry A, Brouwer-Visser J. Early clearance of circulating tumor DNA and association with odronextamab response in relapsed/refractory FL and DLBCL. Blood Adv. 2025 Dec 9;9(23):6130-6140. doi: 10.1182/bloodadvances.2025016332. PMID 40902079
- [Derived] Danilov AV, Kambhampati Thiruvengadam S, Linton K, Cumings K, Chirikov V, Mutebi A, Bains Chawla S, Chhibber A, Rivas Navarro F, Marques Goncalves F, Wang A, Ding Z, Alshreef A, Favaro E, Hoehn D, Sureda A. Indirect comparison of epcoritamab vs chemoimmunotherapy, mosunetuzumab, or odronextamab in follicular lymphoma. Blood Adv. 2025 Aug 12;9(15):3754-3765. doi: 10.1182/bloodadvances.2024015274. PMID 40472301
- [Derived] Kim WS, Kim TM, Cho SG, Jarque I, Iskierka-Jazdzewska E, Poon LM, Prince HM, Zhang H, Cao J, Zhang M, Tessoulin B, Oh SY, Lim F, Carpio C, Tan TD, Ayyappan S, Gutierrez A, Cai J, Ufkin M, Shariff S, Brouwer-Visser J, Chaudhry A, Mohamed H, Ambati S, Walewski J; ELM-2 Investigators. Odronextamab monotherapy in patients with relapsed/refractory diffuse large B cell lymphoma: primary efficacy and safety analysis in phase 2 ELM-2 trial. Nat Cancer. 2025 Mar;6(3):528-539. doi: 10.1038/s43018-025-00921-6. Epub 2025 Mar 17. PMID 40097657
- See also: Related Info — https://elmclinicalresearchstudies.com/